CLINICAL TRIAL: NCT00000215
Title: IV Cocaine Abuse: A Laboratory Model
Brief Title: IV Cocaine Abuse: A Laboratory Model - 4
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Collaborators: Columbia University (Other)
Purpose: Treatment
Other Study IDs: NIDA-06234-4; R01-06234-4
Record Dates: First submitted 1999-09-20; First posted 1999-09-21 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2016-10

CONDITIONS: Cocaine-Related Disorders
Keywords: cocaine dependence
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Pergolide

INTERVENTIONS:
Drug: Pergolide

SUMMARY:
The purpose of this study is to evaluate the effects of pergolide on cocaine taking and on the physiological and subjective effects of cocaine, including cocaine craving in non-opiate dependent cocaine users.

ELIGIBILITY:
Please contact site for information.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0
Dates: Study Completion 2001-12

PRIMARY OUTCOMES:
Direct cocaine effects (cardio, subjective)
Interaction of cocaine/pergolide on cardio
Interaction of coc/pergolide on coc's subjective
Effects of pergolide on cocaine craving

CONTACTS AND LOCATIONS:
Overall Officials: Richard Foltin, Ph.D., Principal Investigator — Columbia University
Locations (1):
- Columbia University, New York, New York, United States